CLINICAL TRIAL: NCT03745027
Title: Follicular Fluid Sialic Acid Levels in in Vitro Fertilization Cycles
Brief Title: Follicular Fluid Sialic Acid Levels in IVF Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014.1.1
Record Dates: First submitted 2018-11-10; First posted 2018-11-19 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-11

CONDITIONS: in Vitro Fertilization
Keywords: in vitro fertilization; sialic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In vitro fertilization (Experimental): Paients undergoing in vitro fertilization with Gonadotropin-releasing Hormone agonist. Follicular fluid sialic acid levels will be measured.
  Interventions: Diagnostic Test: in vitro fertilization

INTERVENTIONS:
Diagnostic Test: in vitro fertilization — All patients underwent gonadotropin-releasing hormone agonist (GnRHa) treatment for in vitro fertilization and Follicular fluid sialic acid levels are measured.

SUMMARY:
This cross-sectional study was conducted at the Reproductive Endocrinology and Invitro Fertilization (REI) unit of our hospital, following the approval of the hospital's ethics committee. Patients who underwent gonadotropin-releasing hormone agonist (GnRHa) treatment were enrolled in the study. During oocyte retrieval, follicular fluids of mature follicles (≥18 mm) were collected and pooled for each patient. The thiobarbituric acid method was used for the sialic acid levels and the absorbance values were measured by a spectrophotometer at 549 nm.

DETAILED DESCRIPTION:
This cross-sectional study was conducted at the Reproductive Endocrinology and Invitro Fertilization (REI) unit our hospital, following the approval of the hospital's ethics committee. The inclusion criteria were as follows; under 40 years of age, normal thyroid and prolactin hormone levels, a basal follicle stimulating hormone (FSH) level <10 mIU/mL, BMI of 19-30 kg/m2. Exclusion criteria: a history of ovarian surgery, endometriosis, uterine anomaly, any endocrine disease including congenital adrenal hyperplasia, smokers, use of any medications and hormones in the last 3 months. Before the IVF treatment serum follicle stimulating hormone (FSH), luteinizing hormone (LH), prolactin (PRL), thyroid-stimulating hormone (TSH), and estradiol (E2) levels were measured on the third day of the cycle. Age, body mass index, duration of stimulation, duration of infertility, the total dose of gonadotropins, E2 on the day of hCG administration, number of oocytes retrieved, fertilization rate, and pregnancy rate were recorded.

All patients underwent gonadotropin-releasing hormone agonist (GnRHa) treatment. Oocyte retrieval was done 36 hours after the hCG injection and ICSI was used for all patients. Embryo transfer was performed 48-72 hours after the oocyte retrieval.

During oocyte retrieval, follicular fluids of mature follicles (≥18 mm) were collected from the first follicle entered and were aspirated for each patient. Follicle aspirates, which were not clear and contaminated with blood, were excluded. Total and free sialic acid levels were measured in the follicular fluid.

ELIGIBILITY:
Inclusion Criteria:

* under 40 years of age,
* normal thyroid and prolactin hormone levels,
* a basal follicle stimulating hormone (FSH) level <10 mIU/mL,
* body mass index (BMI) of 19-30 kg/m2

Exclusion Criteria:

* a history of ovarian surgery, endometriosis, uterine anomaly,
* any endocrine disease including congenital adrenal hyperplasia,
* smokers,
* use of any medications and hormones in the last 3 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who become pregnant | during procedure
  Number of patients who become pregnant will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan A Çetin, Principal Investigator — KSSTRH
Locations (1):
- Kanuni SSRTH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided